CLINICAL TRIAL: NCT00551824
Title: Evaluation of Topical Mitomycin C as Adjuvant Drug to Endoscopic Esophageal Dilation in Children
Brief Title: Evaluation of Topical Mitomycin C as Adjuvant Drug to Esophageal Dilation in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MITOMYCIN
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2008-04-09 (Estimated); Status verified 2007-10

CONDITIONS: Esophageal Stricture; Caustic Esophageal Stricture; Peptic Esophageal Stricture; Post-Surgical Esophageal Stricture
Keywords: esophageal stricture
MeSH Terms: conditions — Esophageal Stenosis | interventions — Mitomycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): First dilation session with topical mitomycin applied over esophageal mucosa after dilation.
  Second dilation session (after 14 days): standard dilation without topical mitomycin.
  Interventions: Drug: Mitomycin C
- 2 (Experimental): First dilation session: standard dilation without topical mitomycin.
  Second dilation session (after 14 days) with topical mitomycin applied over esophageal mucosa after dilation.
  Interventions: Drug: Mitomycin C

INTERVENTIONS:
Drug: Mitomycin C — Esophageal dilation session with topical mitomycin applied over esophageal mucosa after dilation.

SUMMARY:
This study aims to evaluate mitomycin C as an adjunct to endoscopic treatment of esophageal strictures.

This is a crossover, controlled, clinical trial in which children with esophageal stricture will be randomized in two groups to receive either topical mitomycin or no additional treatment during standard esophageal dilation session.

DETAILED DESCRIPTION:
Topical mitomycin C has been used as an adjunct drug to endoscopic treatment of aero-digestive strictures. There has been some case reports and case series of this application in esophageal strictures in children, with good results. Nevertheless, it lacks a controlled clinical trial to access the efficacy of the mitomycin C in this context.

This study aims to evaluate mitomycin C as an adjunct to endoscopic treatment of esophageal strictures.

This is a crossover placebo-controlled single-blind clinical trial.

Patients: Subjects up to 18 year-old, with esophageal stricture requiring endoscopic dilation, either due to dysphagia or by stricture preventing passage of the endoscope.

Inclusion criteria:

* peptic esophageal stricture
* post-surgical esophageal stricture
* caustic esophageal stricture

The patient will be randomized by one treatment group, either A or B.

* A. during the first endoscopic procedure it will be applied of topical mitomycin C over the esophageal mucosa after dilation, then the second procedure (in two weeks) will be performed as a standard dilation, without mitomycin C.
* B. the first procedure will be performed in a standard way, and after two weeks, in the second procedure mytomicin-C will be spread over the esophageal mucosa.

The allocation will not be informed to the patient. At the end of the study protocol, the patients will be clinically evaluated and the dilation program will continue on discretion of the assistant doctor. The target esophageal bore is 11 mm (or 12.8 mm if age above 5 yrs).

Mitomycin C will be applied over the esophageal mucosa in the site of stricture after dilation with a cotton pledget soaked in solution (0.4mg/ml) by three minutes. The pledget will he held over the mucosa with a biopsy forceps.

Clinical evaluation. Dysphagia will be evaluated by a structured questionnaire, using a Likert scale. The patient will answer the questionnaire daily.

Main outcome measure: Number of days with improved symptom (dysphagia) after a session.

ELIGIBILITY:
Inclusion Criteria:

* children with esophageal strictures
* and dysphagia
* or stricture preventing endoscope to pass over it.

Exclusion Criteria:

* congenital esophageal stricture
* stricture associated to eosinophilic esophagitis

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-12 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Number of days with improved symptom (dysphagia) after dilation session. | 14 days

SECONDARY OUTCOMES:
Esophageal diameter | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo S Machado, PhD, Principal Investigator — Disciplina de Gastroenterologia Pediátrica, UNIFESP/EPM
Locations (1):
- Hospital São Paulo, São Paulo, São Paulo, Brazil